CLINICAL TRIAL: NCT05810896
Title: Improving Outpatient Comprehensive Atrial Fibrillation Care Across Central North Carolina Through Direct Primary Care and Patient Engagement
Brief Title: AF at Home: A Virtual Education Program for Patients With Atrial Fibrillation (AF)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); Wake Forest University (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-1350b
Record Dates: First submitted 2023-03-30; First posted 2023-04-13 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Investigators will use a pre-test post-test model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AF at Home (Experimental): All recruited participants will participate in the AF at Home educational intervention.
  Interventions: Other: AF at Home

INTERVENTIONS:
Other: AF at Home — The AF at Home education program will be delivered via Zoom videoconferencing technology and will include 6, 1-hour long sessions that involve education on AF self-monitoring and self-management. Each session will include a didactic presentation and open Q&A. Supplementary educations materials will be made available to participants.

SUMMARY:
The goal of this study is to determine the effectiveness of a direct-to-patient virtual education program ("AF at Home") for adults with atrial fibrillation (AF). The main questions this study aims to answer are:

1. Will participants in the educational program have improvement in quality of life, self-monitoring, and self-management strategies after program completion?
2. Will patient level quality of AF care improve for participants in the educational program?

Participants will be asked to:

* Participate in six hours of virtual education sessions over three weeks via Zoom.
* Complete online questionnaires before the program starts and after its completion.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosis of non-valvular or valvular atrial fibrillation
* Age >/= 18

Exclusion Criteria:

* Unable to provide informed consent
* Incarcerated patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change Atrial Fibrillation Effect on Quality-of-life Questionnaire (AFEQT) Score | Baseline and 3 weeks
  The AFEQT questionnaire is a validated tool used to measure self-reported quality of life specifically for patients with atrial fibrillation. The questionnaire includes 20 questions measured on a 7-point Likert scale (1= not at all to 7=extremely) with 3 subcategories. The subcategories include symptoms (questions 1-4), daily activities (questions 5-12), and treatment concerns (questions 13-18). Scoring provides an overall AFEQT score (based on questions 1-18), and a treatment satisfaction score (based on questions 19-20). Treatment satisfaction scores are not included in the overall AFEQT score. Overall or subcategory scores range from 0-100. A score of 100 corresponds to no disability, and a score of 0 corresponds to total disability.

SECONDARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System 29 (PROMIS-29) Global Pain Intensity Scores | Baseline and 3 weeks
  The PROMIS-29 questionnaire measures pain intensity across 7 domains with 4 questions in each domain (physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain interference), and one global pain intensity question. Each domain score ranges from 4-20 with higher scores indicating more of the symptom being measured. Global pain intensity score ranges from 0-10 (0-no pain to 10=highest pain level).
Change in Cardiac Anxiety Questionnaire (CAQ) | Baseline and 3 weeks
  The CAQ is a self-reported measure that assesses anxiety related specifically to cardiac symptoms. The CAQ contains 18 questions rated on a 5-point Likert scale (0=never to 4=always). The questionnaire contains 3 subcategories including fear (8 questions), avoidance (5 questions), and attention (5 questions). The higher the score, the more symptoms and or frequency.
Number of Patients Prescribed Appropriate Anticoagulation | Baseline and 1-year post intervention session 6
  This outcome measures the Number of patients prescribed appropriate anticoagulation medication based on risk factors for stroke including congestive heart failure (C), hypertension (H), Age >74 (A2), Diabetes (D), prior stroke or transient ischemic attack (TIA) (S2), vascular disease (V), age 65-74 (A), female sex (Sc), commonly referred to as CHA2DS2-VASc stroke risk score for patients with atrial fibrillation. CHA2DS2-VASc score includes 7 indicators of stroke risk (age (<65=0, 65-74=1, 75+= 2), sex (male=0, female=1), heart failure (no=0, yes=1), hypertension (no=0, yes=1), prior stroke/TIA (no=0, yes=2), history of vascular disease (no=0, yes=1), and diabetes (no=0, yes=1). Anticoagulation is indicated for a female with a score 3 or higher and males with a score of 2 or higher. This information will be collected from electronic health records.
Number of Patients Prescribed Antiplatelet Therapy for AF Stroke Risk Reduction | Baseline and 1-year post intervention session 6
  This outcome will measure the number of patients who were prescribed antiplatelet therapy for atrial fibrillation stroke risk reduction without comorbid vascular disease. This information will be collected from electronic health records.
Number of Patients with Achievement of Blood Pressure at Target | Baseline and 1-year post intervention session 6
  This outcome will measure the number of patients meeting guideline blood pressure target of systolic blood pressure (SBP) <130 mmHg.This information will be collected from electronic health records.
Number of Patients with Achievement of Heart Rate Target | Baseline and 1-year post intervention session 6
  This outcome will measure the number of patients meeting guideline heart rate target of <110 beats per minute (bpm). This information will be collected from electronic health records.
Number of Patients Prescribed Rhythm Controlling Medications | Baseline and 1-year post intervention session 6
  This outcome will measure the number of patients who are prescribed rhythm controlling medications. This information will be collected from electronic health records.
Number of Emergency Department Visits or Hospital Admissions for AF or Stroke (Healthcare Utilization) | Baseline and 1-year post intervention session 6
  This outcome will measure the number of emergency room visits and/or hospital admissions with a primary or secondary diagnosis of atrial fibrillation or stroke. This information will be collected from electronic health records.
Change in Confidence in Atrial Fibrillation Management (CALM) Scale | Baseline and 3 weeks
  The CALM scale is a newly developed tool to assess self-reported confidence in self-management skills for patients with AF. The CALM scale contains 16 questions to indicate the level of confidence in each item on a range of 0-4 (not confident =0, to extremely confident=3). The higher the score, the more confident in self-management skills.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Gehi, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: Deidentified individual data that supports the results will be shared beginning 12 to 36 months following publication.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] January CT, Wann LS, Calkins H, Chen LY, Cigarroa JE, Cleveland JC Jr, Ellinor PT, Ezekowitz MD, Field ME, Furie KL, Heidenreich PA, Murray KT, Shea JB, Tracy CM, Yancy CW. 2019 AHA/ACC/HRS Focused Update of the 2014 AHA/ACC/HRS Guideline for the Management of Patients With Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society in Collaboration With the Society of Thoracic Surgeons. Circulation. 2019 Jul 9;140(2):e125-e151. doi: 10.1161/CIR.0000000000000665. Epub 2019 Jan 28. No abstract available. PMID 30686041
- [Background] Gallagher C, Rowett D, Nyfort-Hansen K, Simmons S, Brooks AG, Moss JR, Middeldorp ME, Hendriks JM, Jones T, Mahajan R, Lau DH, Sanders P. Patient-Centered Educational Resources for Atrial Fibrillation. JACC Clin Electrophysiol. 2019 Oct;5(10):1101-1114. doi: 10.1016/j.jacep.2019.08.007. Epub 2019 Sep 1. PMID 31648734
- [Background] Tripp C, Gehi AK, Rosman L, Anthony S, Sears SF. Measurement of patient confidence in self-management of atrial fibrillation: Initial validation of the Confidence in Atrial fibriLlation Management (CALM) Scale. J Cardiovasc Electrophysiol. 2021 Jun;32(6):1640-1645. doi: 10.1111/jce.15050. Epub 2021 May 12. PMID 33982364
- [Background] Rosman L, Armbruster T, Kyazimzade S, Tugaoen Z, Mazzella AJ, Deyo Z, Walker J, Machineni S, Gehi A. Effect of a virtual self-management intervention for atrial fibrillation during the outbreak of COVID-19. Pacing Clin Electrophysiol. 2021 Mar;44(3):451-461. doi: 10.1111/pace.14188. Epub 2021 Feb 17. PMID 33565642